CLINICAL TRIAL: NCT00033735
Title: Phase III Trial Of Irofulven Vs. 5-Fluorouracil In Patients With Gemcitabine-Refractory Advanced Pancreatic Adenocarcinoma
Brief Title: Irofulven Compared With Fluorouracil in Treating Patients With Pancreatic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069317; MGI-IROF-003; UARIZ-HSC-00305
Record Dates: First submitted 2002-04-09; First posted 2004-01-15 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2012-12

CONDITIONS: Pancreatic Cancer
Keywords: recurrent pancreatic cancer; duct cell adenocarcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Fluorouracil; irofulven

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- fluorouracil (Experimental)
  Interventions: Drug: fluorouracil
- Irofulven (Experimental)
  Interventions: Drug: Irofulven

INTERVENTIONS:
Drug: fluorouracil — 5-fluorouracil will be administered via central venous catheter or PICC beginning at 250mg/m2/ day as continous infusion for a 28 day period.
  Arms: fluorouracil
Drug: Irofulven — Irofulven will be given at 0.55 mg/kg per infusion on Day 1 and and Day 15 every 28 days as a 30 minute iv infusion.
  Arms: Irofulven

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether irofulven is effective in treating pancreatic cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of irofulven with that of fluorouracil in treating patients who have locally advanced or metastatic pancreatic cancer that has not responded to previous treatment with gemcitabine.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare survival of patients with gemcitabine-refractory, advanced pancreatic adenocarcinoma when treated with irofulven vs fluorouracil. II. Compare the objective tumor response rate in patients treated with these regimens. III. Compare the clinical benefit of these regimens as measured by improvement in pain and performance status in these patients.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are randomized 2:1 to irofulven and fluorouracil treatment arms. Arm I: Patients receive irofulven IV over 30 minutes on days 1 and 15. Arm II: Patients receive fluorouracil IV continuously on days 1-28. Courses repeat every 28 days.

PROJECTED ACCRUAL: Approximately 350 patients (233 for arm I and 117 for arm II) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed ductal carcinoma of the exocrine pancreas Locally advanced or metastatic Failed 1, but no more than 1, prior gemcitabine-containing chemotherapy regimen (either as a single agent or in combination with another agent) (See criteria for prior radiation using gemcitabine or fluorouracil at diminished doses in Prior/Concurrent Therapy section) No neuroendocrine or islet cell tumors or lymphoma of the pancreas

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9 g/dL Absolute neutrophil count at least 1,500/mm3 Hepatic: Bilirubin no greater than 2.0 mg/dL AST or ALT no greater than 5.0 times upper limit of normal (ULN) Alkaline phosphatase no greater than 5.0 times ULN Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: No clinically significant active heart disease Other: Fertile patients must use effective contraception No history of retinopathy or macular degeneration No other malignancy within the past 5 years except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix No other significant medical and/or psychiatric condition that would preclude study

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior biologic therapy No concurrent biologic therapy Chemotherapy: See Disease Characteristics At least 21 days since prior chemotherapy and recovered No prior systemic treatment with fluorouracil, fluorouracil-uracil, raltitrexed, or capecitabine in combination with gemcitabine Prior fluorouracil or gemcitabine allowed as radiosensitizing agents when given 2 weeks before, during, or 2 weeks after radiotherapy No prior cumulative mitomycin dose greater than 25 mg/m2 Endocrine therapy: Not specified Radiotherapy: At least 21 days since prior radiotherapy and recovered Surgery: No prior surgery No concurrent surgery Other: At least 21 days since prior participation in other investigational study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2000-01; Primary Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Survival of Irofulven vs. 5-FU | 28 day cycle or until disease progression

SECONDARY OUTCOMES:
Objective Tumor Response of Irofulven vs. 5-FU and Clinical Benefit of Irofulven vs. 5-FU | 28 day cycle or until disease progression

CONTACTS AND LOCATIONS:
Overall Officials: MGI Medical Communications, Study Chair — Eisai Inc.
Locations (1):
- MGI Pharma, Incorporated, Bloomington, Minnesota, United States